CLINICAL TRIAL: NCT04245111
Title: ICG Fluorescence Imaging in Trauma Patients
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Physician, Dartmouth-Hitchcock Medical Center
Other Study IDs: D20027
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Trauma Injury
Keywords: Immunofluorescence; Orthopaedic; Trauma
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open Fracture Cohort: Patients 18 years of age or older. Open extremity fracture. Planned definitive fracture management with external fixation, internal fixation, or joint fusion. Open fracture wound management that includes formal surgical debridement within 72 hours of their injury. Will have all planned fracture care surgeries performed by a participating surgeon or delegate. Provision of informed consent.
  Interventions: Other: Immunofluorescence Imaging
- Complication Cohort: Patients 18 years of age or older. Extremity fracture. Prior definitive fracture management with external fixation, internal fixation, or joint fusion. Superficial, deep, or organ space SSI (as per CDC criteria) at the fracture site that requires operative management. Will have all fracture care surgeries performed by a participating surgeon or delegate. Provision of informed consent
  Interventions: Other: Immunofluorescence Imaging
- Closed Fracture Cohort: Patients 18 years of age or older Closed extremity fracture Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
  Provision of informed consent
  Interventions: Other: Immunofluorescence Imaging

INTERVENTIONS:
Other: Immunofluorescence Imaging — Patients will be administered FDA approved ICG through intravenous injection and imaged by a FDA approved surgical microscope (Pentero or Spy Elite) which is 0.5 meter away from the subject. Both ICG fluorescence and the two imaging systems have been used for routine clinical practice for many years. Figure (a) shows the Schematic sketch of the imaging systems. ICG fluorescence imaging utilizes intravenously injected ICG, which is a fluorescent dye that is FDA-approved for clinical use, illuminated with near-infrared light. The ICG dye is indirectly activated and the dynamic fluorescence due to bone perfusion can be captured by a video rate imaging system.

SUMMARY:
This will be a prospective observational trial to better understand the range and variation associated with bone/soft tissue perfusion in fracture patients and examine the relationship between perfusion, measured using quantitative Indocyanine green (ICG) fluorescence and complications such as surgical site infection (SSI), persistent SSI, and fracture nonunion.

DETAILED DESCRIPTION:
This will be a prospective observational trial to better understand the range and variation associated with bone/soft tissue perfusion in fracture patients and examine the relationship between perfusion, measured using quantitative Indocyanine green (ICG) fluorescence and complications such as surgical site infection (SSI), persistent SSI, and fracture nonunion. Primary outcome measure is complication (either infection, recurrent infection or nonunion). Eligible consenting patients will receive standard of care treatment for their fracture or infection including irrigation and debridement of their operative site and/or fracture fixation. After exposure, 0.1 mg/Kg ICG will be injected intravenously and video rate ICG fluorescence images will be acquired 20 seconds before and 4 minutes after the injection, each before and after debridement. A subset of 38 post-fracture complication patients will undergo surgical treatment for their infection in Center of Innovation Surgery (CIS) and have either an intraoperative Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) after exposure but before the ICG injection or a preoperative DCE-MRI. Patients receiving surgery in the CIS will be required to sign an additional CIS-specific consent document. The need for repeat surgical procedure will be left up to the treating surgeon. If repeat procedure is needed, pre- and post-debridement quantitative ICG fluorescence images will be obtained at each procedure. Study participants will be followed at 2 weeks, 6 weeks, 3 months and 6 months from their index study surgery. Complication including index infection, recurrent infection or delaying union/nonunion will be identified at the time of diagnosis and/or during each participants assessment that occurs during routine outpatient clinic visit. Detailed information on the infection including date of diagnosis, participant signs and symptoms, culture test results, method of treatment(s), and date of resolution will be documented.

4/23/2020: Study recruitment temporarily halted due to COVID-19

ELIGIBILITY:
Inclusion Criteria:

Open Fracture Cohort (Cohort 1)

1. Patients 18 years of age or older.
2. Open extremity fracture.
3. Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Open fracture wound management that includes formal surgical debridement within 72 hours of their injury.
5. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
6. Provision of informed consent.

Established SSI Fracture Cohort (Cohort 2)

1. Patients 18 years of age or older.
2. Extremity fracture.
3. Prior definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Superficial, deep, or organ space SSI (as per CDC criteria) at the fracture site that requires operative management.
5. Will have all fracture care surgeries performed by a participating surgeon or delegate.
6. Provision of informed consent.

Closed Fracture Cohort (Cohort 3)

1. Patients 18 years of age or older.
2. Closed extremity fracture.
3. Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
5. Provision of informed consent.

Exclusion Criteria:

Open Fracture Cohort (Cohort 1)

1. Fracture of the hand.
2. Iodine allergy.
3. Received previous surgical debridement or management of their fracture at a non-participating hospital or clinic.
4. Open fracture managed outside of the participating orthopaedic service.
5. Chronic or acute infection at or near the fracture site at the time of initial fracture surgery.
6. Burns at the fracture site.
7. Incarceration.
8. Expected survival of less than 90 days.
9. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.

Established SSI Fracture Cohort (Cohort 2)

1. Fracture of the hand.
2. Iodine allergy.
3. Received previous surgical debridement to manage the SSI.
4. Incarceration.
5. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.

   Subset: DCE-MRI (Cohort 2-1)
6. the presence of an electronic implant, such as a pacemaker
7. the presence of a metal implant, such as an aneurysm clip
8. the presence of other contraindication(s), as determined by the MRI technologists and radiologists.
9. A history of allergy to iodides
10. A GFR < 30 ml/min as determined by blood test on the day of NIR/MR imaging, or from lab results within 3 months of DCE-MRI for this study

Closed Fracture Cohort (Cohort 3)

1. Fracture of the hand.
2. Iodine allergy.
3. Chronic or acute infection at or near the fracture site at the time of initial fracture surgery.
4. Burns at the fracture site.
5. Incarceration.
6. Expected survival of less than 90 days.
7. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who present with an open fracture will be considered for the open fracture cohort (Cohort 1). Similarly fracture patients who present with an SSI following fracture fixation or joint fusion will be screened for the fracture SSI cohort (Cohort 2). Patients who present with a closed fracture will be considered for the closed fracture cohort (Cohort 3).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Closed Fracture Cohort: Patients 18 years of age or older Closed extremity fracture Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
  Provision of informed consent
  Immunofluorescence Imaging: Patients will be administered FDA approved ICG through intravenous injection and imaged by a FDA approved surgical microscope (Pentero or Spy Elite) which is 0.5 meter away from the subject. Both ICG fluorescence and the two imaging systems have been used for routine clinical practice for many years. Figure (a) shows the Schematic sketch of the imaging systems. ICG fluorescence imaging utilizes intravenously injected ICG, which is a fluorescent dye that is FDA-approved for clinical use, illuminated with near-infrared light. The ICG dye is indirectly activated and the dynamic fluorescence due to bone perfusion can be captured by a video rate imaging system.
Period: Overall Study
Arm/Group | Open Fracture Cohort | Complication Cohort | Closed Fracture Cohort
Started | 13 | 6 | 1
Imaging Completed | 13 | 6 | 1
Completed | 8 (Completed all imaging plus follow up surveys.) | 5 (Completed all imaging plus follow up surveys.) | 0 (Completed all imaging plus follow up surveys.)
Not Completed | 5 | 1 | 1
Not completed — Lost to Follow-up | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Fracture Cohort | Complication Cohort | Closed Fracture Cohort | Total
Number analyzed (Participants) | 13 | 6 | 1 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 5 | 1 | 18
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 42 [23 to 69] | 56 [43 to 74] | 56 [56 to 56] | 47 [23 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5
  Male | 10 | 4 | 1 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 12 | 6 | 1 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 1 | 20
Type of Extremity Fracture [Count of Participants; unit: Participants]
  Open Fracture | 13 | 0 | 0 | 13
  Fracture with Complication | 0 | 6 | 0 | 6
  Closed Fracture | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients That Complete the Protocol
Description: As this is a pilot and feasibility study, the outcome measure is the percent of patients that successfully complete the protocol.
Time Frame: 1 year
Measure: Number; unit: percentage of completed patients
Arm/Group | Open Fracture Cohort | Complication Cohort | Closed Fracture Cohort
Number analyzed (Participants) | 13 | 6 | 1
percentage of completed patients | 61.5 | 83.3 | 0
Statistical Analysis 1: Comparison: Open Fracture Cohort vs Complication Cohort vs Closed Fracture Cohort; No other statistical analysis completed other than percentage of patients completed as reported in the data table section; Test type: Other — No other statistical analysis completed other than percentage of patients completed as reported in the data table section; No other statistical analysis completed other than percentage of patients completed as reported in the data table section

ADVERSE EVENTS:
Time Frame: From enrollment to Study Follow-up completion (12 months post enrollment)
Description: As defined by clinicaltrials.gov
Arm/Group | Open Fracture Cohort | Complication Cohort | Closed Fracture Cohort
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/6 | 0/1
Other Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Fracture Cohort (N=13) | Complication Cohort (N=6) | Closed Fracture Cohort (N=1)
Rehospitalization for procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Rehospitalization for additional planned procedure. Unrelated to study/expected.
Complication due to surgery (General disorders) | 2 (3) | 1 (1) | 0 (0) — complication from surgery post surgical procedure. Unrelated to study/expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT04245111/Prot_SAP_000.pdf